CLINICAL TRIAL: NCT04869930
Title: Establishing a Diagnostic and Therapeutic Index in Autism Spectrum Disorder (ASD) and Fragile X Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nova Mentis Life Science Corp (Industry)
Collaborators: FourthWall Testing (Unknown)
Responsible Party: Sponsor
Other Study IDs: NM101
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Autism Spectrum Disorder; Fra(X) Syndrome
MeSH Terms: conditions — Autism Spectrum Disorder; Fragile X Syndrome | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Autism Spectrum Disorder (ASD): Early childhood (pre-diagnosis) OR existing diagnosis of moderate/severe ASD
  Interventions: Other: specimen collection
- Fragile X Syndrome (FXS): Existing diagnosis of Fragile X Syndrome
  Interventions: Other: specimen collection
- Healthy Controls: No diagnosed chronic conditions
  Interventions: Other: specimen collection

INTERVENTIONS:
Other: specimen collection — participants will submit at minimum two of four required samples: fecal, urine, finger/toe-prick blood, and cheek swab, collected at home via commercially available kits

SUMMARY:
The purpose of this study is to accumulate and quantitatively analyze data on the microbiome, serotonin signaling and genetics, and inflammatory cytokines from patients with Autism Spectrum Disorder and Fragile X Syndrome. Computational analysis of multi-dimensional datasets will be used to establish a "Diagnostic and Therapeutic Index" - an objective set of tools that can help differentiate subtypes of Autism Spectrum Disorder and develop more accurate methods of diagnosis and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Early childhood (pre-diagnosis) OR existing ASD diagnosis (Moderate to Severe)
* Existing FXS diagnosis

Exclusion Criteria:

* Hospitalization
* Enrolled in another clinical study

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Autism Spectrum Disorder (ASD) and Fragile X Syndrome are neurodevelopmental disorders characterized by repetitive behavioral patterns, hypersensitivity, and persistent deficits in social communication. ASD is currently diagnosed exclusively on the basis of neurobehavioral patterning - an approach that (1) cannot distinguish subtle differences between ASD subtypes, (2) is subject to observer bias, and (3) introduces uncertainty regarding root causes and response to treatments. Developmental disorders are often accompanied by various co-occurring medical conditions like gastrointestinal dysfunction or anemia, which can be leveraged to sub-segment the autisms spectrum and improve diagnostics and treatment. Further investigation is needed to define the degree to which specific comorbidities contribute to behavioral symptomology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
microbial diversity profile | 2 years
  genetic analysis of microbial species in fecal samples

SECONDARY OUTCOMES:
differences in serotonin levels | 2 years
  molecular analysis of blood/urine/fecal samples
differential expression of serotonin-related signaling molecules | 2 years
  genetic analysis of cheek swabs

CONTACTS AND LOCATIONS:
Overall Officials: Julia V Perederiy, PhD, Principal Investigator — Nova Mentis Life Science Corp
Locations (1):
- Broward Health Medical Center, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No